CLINICAL TRIAL: NCT01384669
Title: Genetic Expression Alteration Affect on Lateral Neck Node Metastasis of Thyroid Papillary Microcarcinoma : Microarray Analysis
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2011-0212
Record Dates: First submitted 2011-06-27; First posted 2011-06-29 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2013-12

CONDITIONS: Papillary Thyroid Microcarcinoma
MeSH Terms: conditions — Papillary Thyroid Microcarcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — mRNA extract from Thyroid tissue 2mmx2mmx2mm (nomal thyroid and papillary thyroid microcarcinoma >5mm)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: papillary thyroid microcarcinoma without lymph node metastasis
- Group 2: papillary thyroid microcarcinoma with lateral lymph node metastasis

SUMMARY:
In this study, the investigators look at the genetic expressional alteration which influenced on the early lateral neck node metastasis in thyroid papillary microcarcinoma.

DETAILED DESCRIPTION:
Papillary thyroid carcinomas (PTCs) measuring 1.0 cm or less in diameter were defined as papillary thyroid microcarcinomas (PTMCs) by the World Health Organization (WHO), emphasizing on their benign behavior, probably of little clinical significance, which do not affect patients' survival. However, some reported that PTMCs may have aggressive behavior, can cause locoregional recurrences, cervical lymph node metastases, and even distant metastases. But till now, the characteristics of PTMCs with early lateral neck node metastasis were only reviewed and described by the clinicopathological parameters, and no analysis of PTMCs by the gene level is available. In these study, we investigate the genetic expressional alteration which influenced on the early lateral neck node metastasis in thyroid papillary microcarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* age≥20 years old
* Conventional type papillary thyroid microcarcinoma (0.5cm≤tumor size≤1.0cm)
* group 1: no lymph node metastasis /group 2: with lateral neck node metastasis

Exclusion Criteria:

* tumor with capsular invasion (T3 tumor)
* distant metastasis
* combined underlying thyroiditis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who were diagnosed as papillary thyroid microcarcinoma with or without lateral neck node metastasis
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05-26 (Actual); Study Completion 2013-05-26 (Actual)

PRIMARY OUTCOMES:
mRNA expression pattern by microarray analysis | 24-hour after surgical removement
  mRNA expression differences between papillary thyroid microcarcinoma without lateral neck node metastasis and the one with lateral neck node metastasis. (The outcome will be measured within 24-hour after surgical removement using papillary thyroid microcarcinoma tissue.)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Result] Sugitani I, Kasai N, Fujimoto Y, Yanagisawa A. A novel classification system for patients with PTC: addition of the new variables of large (3 cm or greater) nodal metastases and reclassification during the follow-up period. Surgery. 2004 Feb;135(2):139-48. doi: 10.1016/s0039-6060(03)00384-2. PMID 14739848
- [Result] Hedinger C, Williams ED, Sobin LH. The WHO histological classification of thyroid tumors: a commentary on the second edition. Cancer. 1989 Mar 1;63(5):908-11. doi: 10.1002/1097-0142(19890301)63:53.0.co;2-i. PMID 2914297
- [Result] Chow SM, Law SC, Au SK, Mang O, Yau S, Yuen KT, Lau WH. Changes in clinical presentation, management and outcome in 1348 patients with differentiated thyroid carcinoma: experience in a single institute in Hong Kong, 1960-2000. Clin Oncol (R Coll Radiol). 2003 Sep;15(6):329-36. doi: 10.1016/s0936-6555(03)00066-9. PMID 14524486
- [Result] Chow SM, Law SC, Chan JK, Au SK, Yau S, Lau WH. Papillary microcarcinoma of the thyroid-Prognostic significance of lymph node metastasis and multifocality. Cancer. 2003 Jul 1;98(1):31-40. doi: 10.1002/cncr.11442. PMID 12833452
- [Result] Hay ID, Grant CS, van Heerden JA, Goellner JR, Ebersold JR, Bergstralh EJ. Papillary thyroid microcarcinoma: a study of 535 cases observed in a 50-year period. Surgery. 1992 Dec;112(6):1139-46; discussion 1146-7. PMID 1455316
- [Result] Noguchi S, Yamashita H, Murakami N, Nakayama I, Toda M, Kawamoto H. Small carcinomas of the thyroid. A long-term follow-up of 867 patients. Arch Surg. 1996 Feb;131(2):187-91. doi: 10.1001/archsurg.1996.01430140077021. PMID 8611077
- [Result] Yamashita H, Noguchi S, Murakami N, Toda M, Uchino S, Watanabe S, Kawamoto H. Extracapsular invasion of lymph node metastasis. A good indicator of disease recurrence and poor prognosis in patients with thyroid microcarcinoma. Cancer. 1999 Sep 1;86(5):842-9. doi: 10.1002/(sici)1097-0142(19990901)86:53.0.co;2-x. PMID 10463984
- [Result] Wada N, Duh QY, Sugino K, Iwasaki H, Kameyama K, Mimura T, Ito K, Takami H, Takanashi Y. Lymph node metastasis from 259 papillary thyroid microcarcinomas: frequency, pattern of occurrence and recurrence, and optimal strategy for neck dissection. Ann Surg. 2003 Mar;237(3):399-407. doi: 10.1097/01.SLA.0000055273.58908.19. PMID 12616125
- [Result] Lee X, Gao M, Ji Y, Yu Y, Feng Y, Li Y, Zhang Y, Cheng W, Zhao W. Analysis of differential BRAF(V600E) mutational status in high aggressive papillary thyroid microcarcinoma. Ann Surg Oncol. 2009 Feb;16(2):240-5. doi: 10.1245/s10434-008-0233-3. Epub 2008 Nov 26. PMID 19034577
- [Result] Kebebew E, Weng J, Bauer J, Ranvier G, Clark OH, Duh QY, Shibru D, Bastian B, Griffin A. The prevalence and prognostic value of BRAF mutation in thyroid cancer. Ann Surg. 2007 Sep;246(3):466-70; discussion 470-1. doi: 10.1097/SLA.0b013e318148563d. PMID 17717450
- [Result] Rodolico V, Cabibi D, Pizzolanti G, Richiusa P, Gebbia N, Martorana A, Russo A, Amato MC, Galluzzo A, Giordano C. BRAF V600E mutation and p27 kip1 expression in papillary carcinomas of the thyroid <or=1 cm and their paired lymph node metastases. Cancer. 2007 Sep 15;110(6):1218-26. doi: 10.1002/cncr.22912. PMID 17685465
- [Result] Eun YG, Kim SW, Kim YW, Kwon KH. Loss of Raf-1 kinase inhibitor protein expression is associated with lymph node metastasis in papillary thyroid cancer. Otolaryngol Head Neck Surg. 2010 Oct;143(4):544-8. doi: 10.1016/j.otohns.2010.05.025. Epub 2010 Aug 21. PMID 20869566
- [Result] Yin DT, Wang L, Sun J, Yin F, Yan Q, Shen R, He G, Gao JX. Association of the promoter methylation and protein expression of Fragile Histidine Triad (FHIT) gene with the progression of differentiated thyroid carcinoma. Int J Clin Exp Pathol. 2010 May 25;3(5):482-91. PMID 20606729
- [Result] Moses W, Weng J, Khanafshar E, Duh QY, Clark OH, Kebebew E. Multiple genetic alterations in papillary thyroid cancer are associated with younger age at presentation. J Surg Res. 2010 May 15;160(2):179-83. doi: 10.1016/j.jss.2009.05.031. Epub 2009 Jun 17. PMID 19765726
- [Result] Salehian B, Liu Z. Genetic alterations in differentiated thyroid cancers. Endocr Metab Immune Disord Drug Targets. 2009 Sep;9(3):257-68. doi: 10.2174/187153009789044338. Epub 2009 Sep 1. PMID 19594419
- [Result] Ringel MD. Molecular markers of aggressiveness of thyroid cancer. Curr Opin Endocrinol Diabetes Obes. 2009 Oct;16(5):361-6. doi: 10.1097/MED.0b013e32832ff2cb. PMID 19584719
- [Result] Oler G, Camacho CP, Hojaij FC, Michaluart P Jr, Riggins GJ, Cerutti JM. Gene expression profiling of papillary thyroid carcinoma identifies transcripts correlated with BRAF mutational status and lymph node metastasis. Clin Cancer Res. 2008 Aug 1;14(15):4735-42. doi: 10.1158/1078-0432.CCR-07-4372. PMID 18676742
- [Result] Vasko V, Espinosa AV, Scouten W, He H, Auer H, Liyanarachchi S, Larin A, Savchenko V, Francis GL, de la Chapelle A, Saji M, Ringel MD. Gene expression and functional evidence of epithelial-to-mesenchymal transition in papillary thyroid carcinoma invasion. Proc Natl Acad Sci U S A. 2007 Feb 20;104(8):2803-8. doi: 10.1073/pnas.0610733104. Epub 2007 Feb 12. PMID 17296934
- [Result] Yasuoka H, Nakamura Y, Zuo H, Tang W, Takamura Y, Miyauchi A, Nakamura M, Mori I, Kakudo K. VEGF-D expression and lymph vessels play an important role for lymph node metastasis in papillary thyroid carcinoma. Mod Pathol. 2005 Aug;18(8):1127-33. doi: 10.1038/modpathol.3800402. PMID 15803188
- [Result] Zou M, Famulski KS, Parhar RS, Baitei E, Al-Mohanna FA, Farid NR, Shi Y. Microarray analysis of metastasis-associated gene expression profiling in a murine model of thyroid carcinoma pulmonary metastasis: identification of S100A4 (Mts1) gene overexpression as a poor prognostic marker for thyroid carcinoma. J Clin Endocrinol Metab. 2004 Dec;89(12):6146-54. doi: 10.1210/jc.2004-0418. PMID 15579771